CLINICAL TRIAL: NCT02900976
Title: A Pilot Study of Rituximab (RTX) and Third Party Latent Membrane Protein (LMP)-Specific Cytotoxic T-Lymphocytes (LMP-TC) in Pediatric Solid Organ Recipients (SOT) With EBV-Positive CD20-Positive Post-Transplant Lymphoproliferative Disease (PTLD)
Brief Title: Rituximab and LMP-Specific T-Cells in Treating Pediatric Solid Organ Recipients With EBV-Positive, CD20-Positive Post-Transplant Lymphoproliferative Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANHL1522; NCI-2016-01110 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANHL1522; ANHL1522 (Other: Children's Oncology Group); ANHL1522 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2016-09-06; First posted 2016-09-15 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: EBV-Related Post-Transplant Lymphoproliferative Disorder; Monomorphic Post-Transplant Lymphoproliferative Disorder; Polymorphic Post-Transplant Lymphoproliferative Disorder; Recurrent Monomorphic Post-Transplant Lymphoproliferative Disorder; Recurrent Polymorphic Post-Transplant Lymphoproliferative Disorder; Refractory Monomorphic Post-Transplant Lymphoproliferative Disorder; Refractory Polymorphic Post-Transplant Lymphoproliferative Disorder
MeSH Terms: interventions — Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (RTX) (Experimental): Patients with newly diagnosed PTLD who achieve a complete response (CR) after induction receive additional rituximab or biosimilar as in induction.
  Interventions: Biological: Rituximab
- Arm II (LMP-TC) (Experimental): Patients with newly diagnosed PTLD who do not achieve a CR to induction, all relapsed patients after induction, and all patients with refractory disease who received rituximab or biosimilar within 90 days according to institutional guidelines, receive allogeneic LMP1/LMP2-specific cytotoxic T-lymphocytes IV over 1- 2 minutes on days 0 and 7. Cycle continues for up to 42 days in the absence of disease progression or unacceptable toxicity. Patients with PR or SD after first cycle of cycle allogeneic LMP1/LMP2-specific cytotoxic T-lymphocytes receive an additional cycle.
  Interventions: Biological: Allogeneic LMP1/LMP2-Specific Cytotoxic T-Lymphocytes; Biological: Rituximab

INTERVENTIONS:
Biological: Allogeneic LMP1/LMP2-Specific Cytotoxic T-Lymphocytes — Given IV
  Arms: Arm II (LMP-TC)
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima

SUMMARY:
This pilot phase II trial studies how well rituximab and latent membrane protein (LMP)-specific T-cells work in treating pediatric solid organ recipients with Epstein-Barr virus-positive, cluster of differentiation (CD)20-positive post-transplant lymphoproliferative disorder. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. LMP-specific T-cells are special immune system cells trained to recognize proteins found on post-transplant lymphoproliferative disorder tumor cells if they are infected with Epstein-Barr virus. Giving rituximab and LMP-specific T-cells may work better in treating pediatric organ recipients with post-transplant lymphoproliferative disorder than rituximab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of treating pediatric and young adult solid organ transplant recipients who have newly diagnosed, relapsed or refractory Epstein-Barr virus (EBV)-positive CD20-positive post-transplant lymphoproliferative disease (PTLD) with a novel T-cell therapeutic, allogeneic LMP1/LMP2-specific cytotoxic T-lymphocytes (third party latent membrane protein [(LMP]-)]-specific T cells), in a cooperative group setting.

SECONDARY OBJECTIVES:

I. To determine the percentage of eligible patients for whom a suitable LMP-specific T-cell product derived from a third party LMP-specific T-cell bank is available.

II. To estimate the response rate (RR) to three doses of rituximab (RTX) as single agent in children and young adults with newly diagnosed or relapsed EBV-positive CD20-positive PTLD after solid organ transplantation (SOT).

III. To estimate the 2-year event-free survival (EFS) of children and young adults with newly diagnosed, refractory or relapsed EBV-positive CD20-positive PTLD after SOT treated with RTX and/or LMP-specific T cells.

IV. To estimate overall survival (OS) of children and young adults with newly diagnosed, refractory or relapsed EBV-positive CD20-positive PTLD after SOT treated with RTX and/or LMP-specific T cells.

V. To estimate the RR to LMP-specific T cells of newly diagnosed (without complete response to course RTX1), refractory, and relapsed children and young adults with EBV-positive CD20-positive PTLD.

VI. To estimate progression-free survival (PFS) of children and young adults with newly diagnosed, refractory or relapsed EBV-positive CD20-positive PTLD after SOT treated with RTX and/or LMP-specific T cells.

VII. To describe the toxicity of third party LMP-specific T cells in children and young adults with newly diagnosed, refractory or relapsed EBV-positive CD20-positive PTLD after SOT treated with RTX and/or LMP-specific T cells.

VIII. To validate that absence of EBV viremia correlates with RR, EFS and OS.

EXPLORATORY OBJECTIVES:

I. To determine whether third party LMP-specific T cells promote autologous immune reconstitution of EBV-specific T cells.

II. To determine whether EBV viremia is inversely correlated with an increase in EBV-specific T cells in vivo.

III. To determine whether plasma cytokine profile and changes in cytokines over time correlate with treatment response or toxicity (e.g. cytokine release syndrome).

OUTLINE:

INDUCTION (Cohorts A and B): Patients receive rituximab or biosimilar intravenously (IV) on days 1, 8, 15. Cycle continues for up to 21 days in the absence of disease progression or unacceptable toxicity.

Patients are assigned to 1 of 2 arms.

ARM I (RTX, Cohorts A): Patients with newly diagnosed PTLD who achieve a complete response (CR) after induction receive additional rituximab or biosimilar as in induction.

ARM II (LMP-TC, Cohorts A, B, C): Patients with newly diagnosed PTLD who do not achieve a CR to induction, all relapsed patients after induction, and all patients with refractory disease who received rituximab or biosimilar within 90 days according to institutional guidelines, receive allogeneic LMP1/LMP2-specific cytotoxic T-lymphocytes IV over 1- 2 minutes on days 0 and 7. Cycle continues for up to 42 days in the absence of disease progression or unacceptable toxicity. Patients with PR or SD after first cycle of cycle allogeneic LMP1/LMP2-specific cytotoxic T-lymphocytes receive an additional course.

After completion of study treatment, patients are followed up at 1, 2, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a history of solid organ transplantation
* Patients must have biopsy-proven newly diagnosed, relapsed or refractory polymorphic or monomorphic PTLD using the World Health Organization (WHO) classification and that is:

  * CD20 positive
  * EBV positive by Epstein-Barr virus early ribonucleic acid (RNA) (EBER) in situ hybridization (preferred) and/or LMP immunoperoxidase staining
* There must be evaluable disease at study entry either by imaging or by serial endoscopic biopsies.

  * Note: a measurable node must have an LDi (longest diameter) greater than 1.5 cm; a measurable extranodal lesion should have an LDi greater than 1.0 cm; all tumor measurements must be recorded in millimeters (or decimal fractions of centimeters)
* Patients must be considered medically refractory to decreased immunosuppression (50% or greater reduction) for at least 1 week or there must be documentation in the medical chart that decreased immunosuppression would be associated with an unacceptable risk of rejection
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0 or 1

  * Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Myelosuppressive chemotherapy: must not have received within 2 weeks of entry onto this study
* COHORT A and B: Patient must not have received therapy with anti-CD20 monoclonal antibodies within 90 days of entry onto this study
* COHORT C: Patient must have received rituximab at 375 mg/m^2 weekly for at least 3 doses within the last 90 days prior to study enrollment
* Must not have received any prior radiation to any sites of measurable disease
* Must not have received any prior stem cell transplant
* Must not have received investigational therapy within 30 days of entry onto this study
* Must not have received prior EBV or LMP-specific T cells within 90 days of entry onto this study
* Must not have received alemtuzumab or other anti-T-cell antibody therapy within 28 days of entry onto this study
* COHORT C: HLA typing is available and will be submitted at the time of enrollment.

Exclusion Criteria:

* Burkitt morphology
* Central nervous system (CNS) involvement; CNS status must be confirmed by lumbar puncture

  * Note: lumbar puncture can be performed at the time of diagnosis and does not need to be repeated unless there is a change in neurological status or it was performed more than 14 days prior to study entry
* Bone marrow involvement (> 25%)

  * Note: bone marrow aspiration/biopsy can be performed at the time of diagnosis and does not need to be repeated unless there is a change in peripheral blood counts or it was performed more than 14 days prior to study entry
* Fulminant PTLD defined as: fever > 38 degrees Celsius (C), hypotension, and evidence of multi-organ involvement/failure including two or more of the following:

  * Bone marrow (including pancytopenia without any detectable B-cell proliferation)
  * Liver (coagulopathy, transaminitis and/or hyperbilirubinemia)
  * Lungs (interstitial pneumonitis with or without pleural effusions)
  * Gastrointestinal hemorrhage
* Any documented donor-derived PTLD
* Hepatitis B or C serologies consistent with past or current infections because of the risk of reactivation with rituximab
* Severe and/or symptomatic refractory concurrent infection other than EBV
* Pregnant females are ineligible since there is no available information regarding human fetal or teratogenic toxicities
* Lactating females are not eligible unless they have agreed not to breastfeed their infants
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation and for 12 months following completion of study therapy.
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2025-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte Wistinghausen, Principal Investigator — Children's Oncology Group
Locations (38):
- United States (38):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Wistinghausen B, Toner K, Barkauskas DA, Jerkins LP, Kinoshita H, Chansky P, Pezzella G, Saguilig L, Hayashi RJ, Abhyankar H, Scull B, Karri V, Tanna J, Hanley P, Hermiston ML, Allen CE, Bollard CM. Durable immunity to EBV after rituximab and third-party LMP-specific T cells: a Children's Oncology Group study. Blood Adv. 2024 Mar 12;8(5):1116-1127. doi: 10.1182/bloodadvances.2023010832. PMID 38163318

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (RTX) | Arm II (LMP-TC)
Started | 2 | 16
Completed | 2 | 7
Not Completed | 0 | 9
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Progressive disease | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (RTX) | Arm II (LMP-TC) | Total
Number analyzed (Participants) | 2 | 16 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 14 | 16
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6 (7.1) | 10.1 (6.4) | 9.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 0 | 10 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 1 | 11 | 12
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 1 | 8 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 16 | 18

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Assigned to Arm Latent Membrane Protein-specific T-cells (LMP-TC) With Successful LMP-specific T Cell Product Match, Were Treated Within Two Weeks of the Expected Start Date, and Received Both Weekly Doses
Description: The percentage of patients assigned to Arm LMP-TC who had a suitable LMP-specific T-cell product, were treated within two weeks of the expected start date, and received both weekly doses in a cooperative multi-institutional setting. A statistical analysis was planned, but not performed because accrual was stopped early and the sample size required for the analysis was not reached.
Time Frame: Day 8 of the first LMP-TC cycle (cycle = 42 days)
Population: 2 Arm I (RTX) patients and 1 Arm II (LMP-TC) patient who came off protocol therapy prior to Callback were excluded from this analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm II (LMP-TC)
Number analyzed (Participants) | 15
Percentage of patients | 86.7 [59.5 to 98.3]

2. Secondary Outcome: Percentage of Patients Successfully Matched to a Latent Membrane Protein (LMP)-Specific T Cell Product Derived From a Third Party LMP-specific T Cell Bank
Description: Will be assessed using an exact one-sided binomial 95% confidence interval to get a lower bound for the actual rate.
Time Frame: Day 1 of the first LMP-TC cycle (cycle = 42 days)
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival
Description: Will be assessed using Kaplan-Meier estimates, for all patients combined and separately for each cohort.
Time Frame: Time to first occurrence of progression or death (events) or loss to follow-up or survival to analysis date (non-events), assessed 12 months from enrollment of the last patient on the study
Reporting Status: Not Posted

4. Secondary Outcome: Event-free Survival (EFS)
Description: Will be assessed using Kaplan-Meier estimates, for all patients combined and separately for each cohort.
Time Frame: as for outcome 3
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival (OS)
Description: Will be assessed using Kaplan-Meier estimates, for all patients combined and separately for each cohort.
Time Frame: as for outcome 3
Reporting Status: Not Posted

6. Secondary Outcome: Response Rate (RR) to Rituximab
Description: Will be assessed using exact two-sided binomial 95% confidence intervals to get estimates of the response rate. Will be evaluated in Cohorts A and B only (combined and separately).
Time Frame: Up to week 3
Reporting Status: Not Posted

7. Secondary Outcome: Response Rate (RR) to LMP-specific T Cells
Description: Will be assessed using exact two-sided binomial 95% confidence intervals to get estimates of the response rate. Will be evaluated in all Cohorts combined and in each Cohort separately.
Time Frame: Up to week 6
Reporting Status: Not Posted

8. Secondary Outcome: Absence of Epstein-Barr Virus Viremia
Description: Will be correlated with response rate (RR), event-free survival (EFS) and overall survival (OS). Using the log-rank test for EFS and OS and the exact conditional test of proportions (Fisher's exact test for RR, both for all patients combined and stratified by cohort.
Time Frame: Up to 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Toxicities will be described using descriptive statistics. Toxicity monitoring and analysis will be performed based on "as treated".
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Enrollment up to 5 years after enrollment
Description: The SAE table reflects NCI CTCAEs submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Not every patient from Arm LMPTC received induction therapy (refractory patients are excluded), so the denominator for Arm LMPTC Induction is less than the denominator for Arm LMPTC
Groups:
- Arm I (RTX) Induction; Arm II (LMP-TC) Induction: Patients receive rituximab or biosimilar intravenously (IV) on days 1, 8, 15. Cycle continues for up to 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm I (RTX) Induction | Arm II (LMP-TC) Induction | Arm I (RTX) | Arm II (LMP-TC)
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/11 | 0/2 | 3/15
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/11 | 0/2 | 6/15
Other Adverse Events (participants affected / at risk) | 2/2 | 5/11 | 1/2 | 3/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (RTX) Induction (N=2) | Arm II (LMP-TC) Induction (N=11) | Arm I (RTX) (N=2) | Arm II (LMP-TC) (N=15)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 0 | 3
Death NOS (General disorders) | 0 | 0 | 0 | 2
Fever (General disorders) | 0 | 0 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 3
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (RTX) Induction (N=2) | Arm II (LMP-TC) Induction (N=11) | Arm I (RTX) (N=2) | Arm II (LMP-TC) (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 4 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0 | 1
White blood cell decreased (Investigations) | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/76/NCT02900976/Prot_SAP_000.pdf